CLINICAL TRIAL: NCT06704295
Title: High Impact E-cigarette Advertisement Features
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Julia Chen-Sankey, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2024002290; R00CA242589 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Vaping Behavior
Keywords: E-cigarette advertisement; Vaping; Complete switching; Cigarette smoking cessation; Young adults; E-cigarette marketing; Tobacco policy
MeSH Terms: conditions — Vaping; Tobacco Use Cessation | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Control ad: Dark gray product with tobacco flavor name (Other)
  Interventions: Behavioral: Control ad with dark gray product with tobacco flavor name
- Dark gray product with strawberry flavor name (Experimental)
  Interventions: Behavioral: Dark gray product with strawberry flavor name
- Colorful (strawberry color) product with strawberry flavor name (Experimental)
  Interventions: Behavioral: Colorful (strawberry color) product with strawberry flavor name
- Colorful (strawberry color) product with strawberry flavor name and strawberry image (Experimental)
  Interventions: Behavioral: Colorful (strawberry color) product with strawberry flavor name and image
- Colorful (strawberry color) product with strawberry flavor features (Experimental): Colorful (strawberry color) product with strawberry flavor name + strawberry image + strawberry flavor sensation descriptor
  Interventions: Behavioral: Colorful (strawberry color) product with strawberry flavor features
- Colorful (strawberry color) product with strawberry flavor features and choice claim (Experimental): Colorful (strawberry color) product with strawberry flavor name + strawberry image + strawberry flavor sensation descriptor + flavor choice claim
  Interventions: Behavioral: Colorful (strawberry color) product with strawberry flavor features and choice claim

INTERVENTIONS:
Behavioral: Control ad with dark gray product with tobacco flavor name — The e-cigarette ad with a dark gray product with a tobacco flavor name
  Arms: Control ad: Dark gray product with tobacco flavor name
Behavioral: Dark gray product with strawberry flavor name — The e-cigarette ad with a dark gray product with a strawberry flavor name
  Arms: Dark gray product with strawberry flavor name
Behavioral: Colorful (strawberry color) product with strawberry flavor name — The e-cigarette ad with a colorful (strawberry color) product with strawberry flavor name
  Arms: Colorful (strawberry color) product with strawberry flavor name
Behavioral: Colorful (strawberry color) product with strawberry flavor name and image — The e-cigarette ad with colorful (strawberry color) product with strawberry flavor name and strawberry image
  Arms: Colorful (strawberry color) product with strawberry flavor name and strawberry image
Behavioral: Colorful (strawberry color) product with strawberry flavor features — The e-cigarette advertisement with colorful (strawberry color) product with strawberry flavor name, strawberry image, and strawberry flavor sensation descriptor
  Arms: Colorful (strawberry color) product with strawberry flavor features
Behavioral: Colorful (strawberry color) product with strawberry flavor features and choice claim — The e-cigarette ad with colorful (strawberry color) product with strawberry flavor name, strawberry image, strawberry flavor sensation descriptor, and flavor choice claim
  Arms: Colorful (strawberry color) product with strawberry flavor features and choice claim

SUMMARY:
This randomized controlled trial aims to examine the effects of high-impact e-cigarette advertisement features among young adults of various tobacco-use statuses. Previous research on examining the effects of e-cigarette advertisement features found that flavor-related features (e.g., flavor-associated product color, name and image, flavor sensation descriptor, and flavor choice claim) may have the largest impact on shaping young adults' perceptions and use intentions of e-cigarettes. No research so far has solely focused on examining the effects of those high-impact flavor-related advertisement features. The present study assessed the effects of high-impact flavor-related advertisement features, including flavor descriptor name, e-cigarette product color (which indicates flavors), flavor-related image, flavor sensation descriptor, and flavor choice claim on perceptions and behavioral intentions among a large online sample of young adults aged 18-30 who either smoke cigarettes or do not use tobacco products. The study is a six-group RCT with parallel assignments that will be delivered through an online self-administered questionnaire consisting of one session. Participants will be randomly assigned to one of six trial arms: 1) dark gray product with tobacco flavor name, 2) dark gray product with strawberry flavor name, 3) colorful (strawberry color) product with strawberry flavor name, 4) colorful (strawberry color) product with strawberry flavor name and strawberry image, 5) colorful (strawberry color) product with strawberry flavor name, strawberry image, strawberry flavor sensation descriptor, and 6) colorful (strawberry color) product with strawberry flavor name, strawberry image, strawberry flavor sensation descriptor, and flavor choice claim. Participants will be exposed to one advertisement corresponding to the assigned condition, and answer survey questions immediately after message exposure.

DETAILED DESCRIPTION:
The FDA considers the marketing plans of new e-cigarette products for premarket tobacco product application approval. Flavor-related advertisement features may entice young adults who do not use tobacco products to use the products but may also generate complete product switching interests among young adults who smoke cigarettes. This study tested the effects of several high-impact e-cigarette advertisement features related to flavors to inform the FDA's policymaking and public health preventive messages.

Setting: The trial will be an experiment delivered through an online self-administered questionnaire consisting of one session over 20 minutes.

Recruitment: Participants will be recruited from the research company Qualtrics from its research panels.

Informed Consent: Participants will provide online consent prior to taking the survey.

Randomization: After providing informed consent and answering pre-exposure questions, the investigator will use Qualtrics programming to randomize participants into one of the six trial conditions. The randomization will use least fill for the allocation of conditions where if the counts for the conditions were equal, the survey would assign the condition sequentially.

Assessment: Participants will take part in one session (estimated at about 20 mins): participants will answer questions assessing tobacco use status, cigarette smoking quit intentions and attempts (only asked young adults who smoke cigarettes), e-cigarette use, and other tobacco product use. They will then view one e-cigarette advertisement for at least 12 seconds and report immediate outcomes, including perceptions and behavioral intentions related to the e-cigarette product they see in the advertisement.

ELIGIBILITY:
Inclusion Criteria:

* Three groups of young adult subjects will be included in the study. The first group is those who are exclusive cigarette smokers (n=1000), defined as those who have smoked at least 100 cigarettes in their lifetime and have smoked at least one cigarette in the past 30 days but have not used e-cigarettes in the past 30 days. The second group is those who are dual users of cigarettes and e-cigarettes (n=1000). Those in this group have smoked more than 100 cigarettes in their lifetime and have smoked a cigarette and also used an e-cigarette in the past 30 days. The third group is those who are non-tobacco users (n=1000), defined as those who have never used any tobacco product before or have never "regularly" used tobacco products before and are currently not using any tobacco products (in the past 30 days).

Exclusion Criteria:

* Any subjects not meeting the inclusion criteria will be excluded from the study. Individuals will be further excluded if they do not provide consent to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3083 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Intentions of using the e-cigarette | Immediately after exposure
  A single item measuring the intentions of using the e-cigarette shown in the ad. Response options are from 0 (Extremely unlikely ) to 10 (Extremely likely).
Intentions of switching completely to the e-cigarette | Immediately after exposure
  A single item measuring participants' intentions of switching completely to the e-cigarette shown in the ad. Response options are from 0 (Extremely unlikely ) to 10 (Extremely likely). This question is only asked among those who smoke cigarettes.

SECONDARY OUTCOMES:
Intentions of using the e-cigarette compared to cigarettes | Immediately after exposure
  A single item measuring the intentions of using the e-cigarette shown in the ad compared to smoking cigarettes. Response options are from 0 (Much less likely ) to 10 (Much more likely).
Intentions of using the e-cigarette compared to other e-cigarettes | Immediately after exposure
  A single item measuring the intentions of using the e-cigarette shown in the ad compared to using other e-cigarette products. Response options are from 0 (Much less likely ) to 10 (Much more likely).
Ad appeal | Immediately after exposure
  A 3-item scale for those who do not use tobacco, measuring to what extent participants perceive the ad they saw to be appealing, including liking the ad, curious about the product shown in the ad, and interest in using the product shown in the ad. Response options are from 0 (Dislike very much ) to 10 (Like very much) for ad liking and 0 (Strongly disagree) to 10 (Strongly agree) for the other two items. A 4-item scale for those who smoke cigarettes, including the same 3-item scale and an additional single item measuring the agreement on whether the ad makes them want to completely switch to the e-cigarette shown in the ad. Response options are from 0 (Strongly disagree) to 10 (Strongly agree).
Perceived absolute harm of using the e-cigarette | Immediately after exposure
  A single item measuring the participants' perception of having health problems from using the e-cigarette shown in the ad. Response options are from 0 (Extremely unlikely ) to 10 (Extremely likely).
Perceived absolute addictiveness of using the e-cigarette | Immediately after exposure
  A single item measuring the participants' perception of becoming addicted to using the e-cigarette shown in the ad. Response options are from 0 (Extremely unlikely ) to 10 (Extremely likely).

OTHER OUTCOMES:
Sensory appeal of the e-cigarette | Immediately after exposure
  Exploratory outcome: Four items measuring the agreement with the sensory appeal of the e-cigarette shown in the ad: the taste of the e-cigarette would: 1) be harsh, 2) be sweet, 3) be fruity, and 4) have a tobacco taste. Response options are from 0 (Strongly disagree) to 10 (Strongly agree).
Positive expectancy of using the e-cigarette | Immediately after exposure
  Exploratory outcome: A single item measuring the agreement with the positive expectancy (I think I might enjoy, experience pleasure, or feel good using this e-cigarette/vape product) of using the e-cigarette shown in the ad. Response options are from 0 (Strongly disagree) to 10 (Strongly agree).
Negative expectancy of using the e-cigarette | Immediately after exposure
  Exploratory outcome: A single item measuring the agreement with the negative expectancy (I think I might feel bad, sick or embarrassed using this e-cigarette/vape product) of using the e-cigarette shown in the ad. Response options are from 0 (Strongly disagree) to 10 (Strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No